CLINICAL TRIAL: NCT02005185
Title: Is Pediatric Anesthesia Associated With Long-term Hippocampal Dysfunction?
Brief Title: Cognitive Effects of Anesthesia on Children
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Davis (Other); UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Sponsor
Other Study IDs: Anes255HippocampalDysfcn
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Procedures Requiring Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 6-11y/o anesthetized at 0-2y/o for >2hrs: 6-11yr olds anesthetized for more than120 minutes before the age of 2.
- 6-11y/o anesthetized @ 0-2y/o for <30min: 6-11 year olds anesthetized for < 30min before the age of 2.
- 6-11y/o anesthetized at 4-7y/o for >2hrs: 6-11 year olds anesthetized for more than 120 min between the ages of 4-7.
- 6-11 y/o healthy control: 6-11 year olds that have never received general anesthesia.

SUMMARY:
Anesthesia for more than 120 minutes given to children less than 2 years of age without coexisting diseases of the central nervous system or the heart cause long-term impairment of recognition memory.

DETAILED DESCRIPTION:
If the subject enrolls in the study, the child will undergo testing for 1) memory, 2) general brain function (i.e. intelligence testing). The parent will complete 3) a parental assessment of the subject's behavior through a standardized questionnaire.

Initial testing of all case and control participants will include an assessment for neurologic and psychiatric conditions, including attention deficit or learning disorders. In addition, each participant will be assessed by the Wechsler Abbreviated Scale of Intelligence (WASI) and the Child Behavioral Checklist (CBCL), which measures children's psychological well-being, competencies and behavioral/emotional problems.

After explaining the study to your child, we will show your child 80 items on a computer screen with a colored border in either in red, green, blue, or yellow. Following a short break, we will show your child 160 items on the screen. Half of these items were previously displayed and half of these items are new. We will ask your child two or three questions: Have we shown you this item before?How sure are you about your response? Your child will be given the choice of one of three categories: Very sure / halfway sure / not sure. What color was it? This question will only be asked if the answer to question 1 was yes.This portion of the test takes about 30 min. Subjects will then participate in a similar test of picture recognition, but we will ask about the location of the original image instead of the color. Your child will then be given a standardized intelligence test. This takes roughly 45 min to an hour to complete.

Some test participants will partake in a reading portion where the test administrator will read a passage to the participant and the child will say whether or not they recognize a series of phrases. This should take about 20 min to complete. Participants are read a passage and presented with a series of sentences. After listening to the text, they will be informed that some of the sentences they will hear are part of the text, whereas other sentences are new. They will be asked to circle "yes" on their answer sheet when they recognize the sentence as being taken directly from the text, and "no" when they think the sentence was not taken from the text and has not been heard before. It will be emphasized that participants must recognize as old only those sentences that included exactly the same words as the sentences encountered in the text. Participants will also be told that for every "yes" answer they would have to select the option "Remember" if they have a clear memory of their encounter with the sentence in mind, and they can further remember some qualitative and contextual information related to the memory itself, or select the option "Familiar" if they have the feeling that the sentence is part of the text story but they cannot recollect any qualitative detail about the encoding of the sentence.

ELIGIBILITY:
Inclusion Criteria:

* General anesthesia for more than 120 minutes between birth and 2 years of age or between ages 4-7
* General anesthesia for less than 30 minutes before the age of 2.
* Use of volatile anesthetic (sevoflurane, isoflurane, halothane or desflurane) with or without nitrous oxide for maintenance of anesthesia.
* Use of fentanyl or morphine as opioids and midazolam as premedication is acceptable. Propofol used for induction only is acceptable.
* Control subjects must never have been exposed to anesthesia or sedation for any procedure.
* English and Spanish speaking subjects

Exclusion Criteria:

* Use of any other agents such as ketamine, meperidine, barbiturates, etomidate, methoxyflurane, chloral hydrate, methadone or lorazepam.
* Low birth weight (<25th percentile)
* premature birth at <36 weeks
* color blindness
* history of brain disease including head trauma
* presence of congenital heart disease
* any other metabolic disease (i.e. diabetes),cancer, or known genetic syndrome.
* significant low blood pressure during their surgery (<30% of baseline for >5min)
* abnormal temperature (deviation from 36.5 degrees C by >1.5 degree C at any point)
* slow heart rate
* low blood oxygen saturation (<93% for >5min.)
* high arterial carbon dioxide levels (>60mm Hg for >5min.)
* control subjects are excluded for any exposure to anesthesia or sedation

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children currently 6-11 years old who have been anesthetized between ages 0-2 or between ages 4-7 and a matched group of children that did not undergo anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2013-11; Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Examine memory in 6-11 year old children | 2-3 hours/subject
  Assess recognition memory using DPSD model in 6-11 year old children

SECONDARY OUTCOMES:
Additional Neuropsychological evaluations | 2-3 hours/subject
  WASI-2, CBCL, listening/reading comprehension (in 8-11 year olds), digit span

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Sall, M.D., PhD, Principal Investigator — Anesthesiologist, Professor, Researcher
Locations (3):
- United States (3):
  - University of California, Davis Center for Mind and Brain, Davis, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - UCSF, San Francisco, California